CLINICAL TRIAL: NCT06637592
Title: Effects of Windlass Versus Calcaneal Taping on Pain, Flexibility and Lower Extremity Function in Football Player With Plantar Fasciitis.
Brief Title: Effects of Windlass Versus Calcaneal Taping in Football Player With Plantar Fasciitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0407
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Football Players
Keywords: plantar fasciitis; taping
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcaneal taping (Experimental): Calcaneal taping is a method employed to offer assistance and relieve discomfort in the heel and ankle area. Start with a clean surface and apply first tape from lateral malleolus, pulling calcaneus in medial direction and attach to medial malleolus. Apply two more tapes in the same manner going distally. Apply an anchor tape at back of heel.
  Interventions: Other: Calcaneal taping
- Windlass taping (Experimental): Begin by anchoring the tape just above the ball of the foot (metatarsal heads). Tear or cut a strip of tape, approximately 2-3 inches long, and place it horizontally around the foot, securing the starting point. Pull the tape diagonally across the bottom of the foot, aiming to support the arch. The tape should be applied with moderate tension to provide support without causing discomfort. While keeping tension on the tape, extend the big toe (great toe) upward. As the toe extends, the tape should tighten, activating the windlass mechanism and providing additional arch support.
  Interventions: Other: Windlass taping

INTERVENTIONS:
Other: Calcaneal taping — Calcaneal taping is a method employed to offer assistance and relieve discomfort in the heel and ankle area. Start with a clean surface and apply first tape from lateral malleolus, pulling calcaneus in medial direction and attach to medial malleolus. Apply two more tapes in the same manner going distally. Apply an anchor tape at back of heel.
  Arms: Calcaneal taping
Other: Windlass taping — Begin by anchoring the tape just above the ball of the foot (metatarsal heads). Tear or cut a strip of tape, approximately 2-3 inches long, and place it horizontally around the foot, securing the starting point. Pull the tape diagonally across the bottom of the foot, aiming to support the arch. The tape should be applied with moderate tension to provide support without causing discomfort. While keeping tension on the tape, extend the big toe (great toe) upward. As the toe extends, the tape should tighten, activating the windlass mechanism and providing additional arch support.
  Arms: Windlass taping

SUMMARY:
Plantar fasciitis is a prevalent ailment that affects the plantar fascia, a dense tissue strip that spans the underside of the foot, from the heel bone to the toes. Football players are especially susceptible to this ailment because of the sport's high-impact nature, which includes repetitive sprinting, jumping, and quick changes in direction. Taping has been used for many years for various ailments. The purpose of this study is to determine the effects of two taping techniques i.e. windlass taping and calcaneal taping on pain, flexibility and lower extremity function in football players.

DETAILED DESCRIPTION:
The study will be a randomized clinical trial conducted at the Pakistan Sports Board and The Raider's football club over a duration of 10 months after synopsis approval. The required sample size for each group, after accounting for a 10% attrition rate, will be 17. Two study groups will be established: Group A, which will receive calcaneal taping among football players, and Group B, which will receive windlass taping among football players. Nonprobability purposive sampling will be employed. Data will be collected using the Numeric Pain Rating Scale (NPRS), Hubscher maneuver, goniometer, and lower extremity functional scale (LEFS) to assess pain severity, flat foot type flexibility, joint range of motion, and lower limb function, respectively. This comprehensive study aims to contribute valuable insights into the effects of calcaneal and windlass taping on football players.

ELIGIBILITY:
Inclusion Criteria:

* positive windlass test
* Pain can appear after a period of intense training, normally declines with the warm up and reappears at the end of training.
* Intense and acute heel pain localized primarily where plantar fascia attaches to the anterior calcaneus.
* The pain presents on first walking in the morning or after a rest period.

Exclusion Criteria:

* Congenital deformity of ankle and foot.
* History of foot and ankle fracture.
* History of ankle and foot surgery.
* Previous surgery or treatment for plantar fasciitis in the previous 6 months.
* Use of an assistive device for ambulation
* Use of an assistive device for ambulation
* Refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
numeric pain rating scale | 1 week
  This is a self-report assessment where participants evaluate their pain using a number scale. The scale normally spans from 0 to 10, where 0 signifies the absence of pain and 10 signifies the most severe agony imaginable.
hubscher maneuver | 1 week
  It is a method of evaluating the flexibility of a pes planus or flat foot type. The test is performed with the patient weight bearing, with the foot flat on the ground, while the clinician dorsiflexors the hallux and watches for an increasing concavity of the Arches of the foot
calcaneal stance phase angle | 1 week
  it is the sngle between calcaneal bisection and vertical line to floor when patient is standing erect on flat surface.
lower extremity functional scale | 1 week
  The Lower Extremity Functional Scale (LEFS) is a patient-reported instrument used to assess the level of functioning in cases of lower extremity musculoskeletal (MSK) disorders. The LEFS has 20 questions with scores ranging from 0 (severe difficulty/inability to execute activity) to 4 (no difficulties). The overall score can be calculated by adding the points for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, Mphil, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Raiders football club, Lahore, Punjab Province
  - Pakistan sports board, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irfan S, Fiaz M. COMPARISON OF CALCANEAL TAPING AND SHAM TAPING IN SHORT TERM MANAGEMENT OF PAIN IN PLANTAR FASCIITIS; A RANDOMIZED CLINICAL TRIAL. Journal of Health and Rehabilitation Research. 2021;1(2):1-4
- [Background] Welte L, Kelly LA, Kessler SE, Lieberman DE, D'Andrea SE, Lichtwark GA, Rainbow MJ. The extensibility of the plantar fascia influences the windlass mechanism during human running. Proc Biol Sci. 2021 Jan 27;288(1943):20202095. doi: 10.1098/rspb.2020.2095. Epub 2021 Jan 20. PMID 33468002
- [Background] Cobden A, Camurcu Y, Sofu H, Ucpunar H, Duman S, Kocabiyik A. Evaluation of the Association Between Plantar Fasciitis and Hallux Valgus. J Am Podiatr Med Assoc. 2020 Mar 1;110(2):Article_2. doi: 10.7547/17-150. PMID 31714797